CLINICAL TRIAL: NCT00905775
Title: Evaluation of Renal Function and Oxidative Stress in Patients Submitted to Myocardial Revascularization Surgery, With Extracorporeal Circulation, and Anesthesia With Isoflurane or Propofol
Brief Title: Renal Function in Patients Submitted to Myocardial Revascularization Surgery
Status: Terminated | Type: Observational
Why Stopped: Failure of recruitment
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Faculdade de Medicina de Botucatu, UNESP, Botucatu, Brasil (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor
Other Study IDs: upeclin/HC/FMB-Unesp-22
Record Dates: First submitted 2009-04-28; First posted 2009-05-21 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2009-05

CONDITIONS: Coronary Disease
Keywords: Isoflurane;; Propofol; Renal functions tests; Cardiovascular tests; revascularization surgery of the myocardium; extracorporeal circulation
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1 Isoflurane: The first group (G1) will be submitted to inhalational general anesthesia with isoflurane (1 CAM, evaluated by expired concentration of isoflurane)
- 2 Propofol: The second group (G2) to targeted venous general anesthesia controlled with propofol. The targeted concentration of propofol will be kept at the predicted plasma concentration from 1 to 2 µg.ml-1 by means of a Diprifusor® infusion pump. During the interval from 10 minutes preceding ECC initiation to 10 minutes after ECC, the propofol concentration will be increased to 2 or 3 µg.ml-

SUMMARY:
Acute renal insufficiency (ARI) represents a frequent and serious complication in patients submitted to cardiac surgery, and is associated with increases in time of hospitalization, costs, morbidity and mortality. Its incidence varies from 3.5% to 31%. The present study aims to evaluate renal function and oxidative stress in patients submitted to revascularization surgery with extracorporeal circulation (ECC), comparing targeted venous anesthesia controlled with propofol and inhalational anesthesia with isoflurane.

DETAILED DESCRIPTION:
Acute renal insufficiency (ARI) represents a frequent and serious complication in patients submitted to cardiac surgery, and is associated with increases in time of hospitalization, costs, morbidity and mortality. Its incidence varies from 3.5% to 31%. The present study aims to evaluate renal function and oxidative stress in patients submitted to revascularization surgery with ECC, comparing targeted venous anesthesia controlled with propofol and inhalational anesthesia with isoflurane.The study will be conducted at the Botucatu Medical School (FMB) and will analyze 60 patients, divided into two randomized groups, submitted to revascularization surgery of the myocardium with ECC. The researcher responsible for data collection from patients will not have knowledge of the type of anesthesia being delivered to the patient.Blood samples will be collected by central venous access for dosing of troponin I, troponin T, CKMB, MDA, creatinine, urea, albumin and cystatin C.Renal function will be evaluated by serum cystatin C and creatinine and the estimated glomerular filtration rate (GFR). GFR will be measured by means of serum cystatin C (Larsson's formula) and by serum creatinine through the Cockcroft-Gault formula (CG) and by the MDRD formula (Modification of Diet in Renal Disease).Markers of renal tubular function will be dosed in the urine, including: alkaline phosphatase, γ - glutamyltransferase(γ-GT), β 2 microglobulin, creatinine and urinary cystatin C.

ELIGIBILITY:
Inclusion Criteria:

* both sexes,
* aged from 18 to 75 years,
* submitted to revascularization surgery of the myocardium
* extracorporeal circulation,
* who had consented to participation by signing the Terms of Free and Clear Consent.

Exclusion Criteria:

* history of hepatic or renal dysfunction,
* history involving acute myocardial infarct
* patients that made use of vitamin C and E;
* patients presenting other cardiac pathologies (valvular, congenital, corrected or not in the same operational act).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included in present study will be patients of both sexes, aged from 18 to 75 years, submitted to revascularization surgery of the myocardium with the use of extracorporeal circulation, who had consented to participation by signing the Terms of Free and Clear Consent.
  Patients excluded will be those with a history of hepatic or renal dysfunction, or a history involving acute myocardial infarct; patients that made use of vitamin C and E; patients presenting other cardiac pathologies (valvular, congenital, corrected or not in the same operational act).
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro TG Vianna, MD, Principal Investigator — Faculdade de Medicina de Botucatu, Unesp
Locations (2):
- Brazil (2):
  - Faculdade de Medicina de Botucatu, Botucatu, São Paulo
  - Upeclin, Botucatu, São Paulo